CLINICAL TRIAL: NCT06151873
Title: Assessment by Surface Electromyography in Cerebral Palsy Footballers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Alejandro Caña Pino, Principal Investigator, University of Extremadura
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 171123
Record Dates: First submitted 2023-11-20; First posted 2023-11-30 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Assessment, Self; Cerebral Palsy; Technology Addiction
MeSH Terms: conditions — Cerebral Palsy; Technology Addiction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Active Comparator): control group sample, healthy subjects without musculoskeletal, neurological or vestibular disorders may participate.
  Interventions: Diagnostic Test: Adapted sport
- Subjects with neurological damage (Experimental): Subjects with cerebral palsy/acquired brain damage belonging to the Spanish National Soccer Team with cerebral palsy and acquired brain damage may participate as an experimental group.
  Interventions: Diagnostic Test: Adapted sport

INTERVENTIONS:
Diagnostic Test: Adapted sport — control group sample, healthy subjects without musculoskeletal, neurological or vestibular alterations can participate.
  Arms: Healthy subjects
Diagnostic Test: Adapted sport — Subjects with cerebral palsy/acquired brain damage belonging to the Spanish National Soccer Team with cerebral palsy and acquired brain damage may participate as an experimental group.
  Arms: Subjects with neurological damage

SUMMARY:
Adapted sport is constantly evolving thanks to the technological and scientific advances in the field of sports that are being developed in our era. Until a few years ago, the study of training, loads, volumes and work intensities were the focus of attention, but nowadays, expanding towards recovery of the individual and consequently to an improvement of the assessments and treatments from the point of view of the alteration of the movement. Impaired motor control is a consequence of most central nervous system (CNS) movement disorders, such as cerebral palsy. A common physical examination includes assessment of passive muscle elongation endurance, isometric and isotonic testing. This test is used to judge the degree and nature of muscle hyperendurance, to determine etiology at the muscle tissue and/or motor control level, and to infer consequences for overall motor performance in functional tasks. Although this physical examination is in widespread clinical use and provides clinically essential information, it is still a subjective assessment and depends on several factors such as intra- and inter-examiner variability.this variability and subjectivity calls for a consensus on the interpretation and measurement of muscle neurophysiological responses in patients with neurological diseases.Generally, the assessment instruments used for the analysis of hypertonia in adapted sports are based on standardized tests and trials. Specifically, in CP (Cerebral Palsy)-Football, hypertonia is assessed by the degrees of spasticity of the modified Ashworth Scale. There is a need for instrumental assessment to validate subjectivity and thus facilitate the applicability, objectivity, characterization and monitoring of the pathology, such as surface electromyography (EMS).

The tests will be performed in a control group of healthy subjects and an experimental group with subjects belonging to the Spanish National Football Team of cerebral palsy and acquired brain damage. After collecting the records, the behavioral patterns in both groups will be evaluated, establishing possible differences between them for the clinimetric indicators analyzed related to muscle activity, thus allowing a characterization of the sample.

Subsequently, by means of the post-exertion assessment of the experimental group, we will analyze the influence of muscle fatigue after an international soccer match.

Therefore, the development of the project aims to provide clinical health professionals and professionals in sports physical activity with evaluative tools (EMG) sensitive to clinical changes that allow characterizing, classifying and observing the evolution of their athletes through a simple, fast and agile characterization of indicators based on surface electromyography for patients with cerebral palsy and acquired brain damage.

ELIGIBILITY:
Control group

Inclusion Criteria:

* healthy subjects with no musculoskeletal, neurological or vestibular disorders

Exclusion Criteria:

* vestibular, neurological and musculoeskeletal disorders

Experimental group

Inclusion criteria:

- subjects with cerebral palsy/acquired brain damag. FT1, FT2 and FT3 soccer clasification.

Exclusion criteria

- healthy subjects with no musculoskeletal, neurological or vestibular disorders

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Baseline muscle activity | one week
  Recording of muscle activity by surface electromyography at rest or basal state of the spastic musculature used in the international sports classification: calf-soleus; hamstrings; adductors.The unit is microvolts
Isometric muscle activity | one week
  Recording of isometric muscle activity by surface electromyography of the spastic musculature used in international sports classification: calf-soleus; hamstrings; adductors. The unit is microvolts

SECONDARY OUTCOMES:
weight | one week
  Descriptive variable. Its unit of measurement is Kilograms
Height | one week
  Descriptive variable. Its unit of measurement is meters
Age | one week
  Descriptive variable. Its unit of measurement is years
sports classification | one week
  Descriptive variable. Player classification according to disability. The values are FT1, FT2 and FT3, with FT1 being the most disabled players.
Affected hemibody | one week
  Descriptive variable. Affected hemibody. Right, left or both.
Modified Ashworth Scale | one week
  The Modified Ashworth Scale is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Extremadura, Badajoz, Spain